CLINICAL TRIAL: NCT04177927
Title: Does Endtidalcarbondioxide Monitoring in Gastrointestinal Endoscopy Have a Clinical Advantage?
Brief Title: Endtidalcarbondioxide Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, mesure gul nihan ozden, Principal investigator, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 053
Record Dates: First submitted 2019-11-20; First posted 2019-11-26 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Gastrointestinal Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endtidalcarbondioxide monitoring group (Experimental): The patients performed gastrointestinal endoscopy will be monitored with Capnostream 20p / Coviden for etCO2 (End tidal CO2), RR (Respitarory rate), SpO2 and PR (heart rate).
  Interventions: Device: Capnostream 20p / Coviden
- Control Group (Active Comparator): Rutine monitorization will be performed to control group of patients.
  Interventions: Device: Rutine monitoring

INTERVENTIONS:
Device: Capnostream 20p / Coviden — The special nasal canule is used for detection carbondioxide from breathe of patients
  Arms: endtidalcarbondioxide monitoring group
Device: Rutine monitoring — peripheric Oxygen saturation is monitored.
  Arms: Control Group

SUMMARY:
Does Endtidalcarbondioxide Monitoring in Gastrointestinal Endoscopy Have a Clinical Advantage?

DETAILED DESCRIPTION:
This study will be randomized prospectively and conducted in Sancaktepe Prof.Dr. Dr. İlhan Varank Training and Research Hospital Endoscopy Unit. After the approval from institute ethics committee, and obtaining written informed consent, sixty patients with ASA I-II who underwent lumbar spinal surgery between 18 and 65 years of age were included in the study. Patients with existing heart and lung disease, liver and kidney failure, morbidly obese, using psychiatric drugs, having malignancy, pregnant and lactating patients will not be included in the study. All patients admitted to the endoscopy unit will be monitorized for noninvasive arterial blood and BiS (Bispectral Index) monitorization. Some of the patients will undergo standard monitoring HR (heart rate) and SpO2 (peripheral oxygen saturation). Other patients will be placed in appropriate nasal cannula Capnostream 20p / Coviden for etCO2 (End tidal CO2), RR (Respitarory rate), SpO2 and PR (heart rate) monitorization. Prior to endoscopic intervention, fentanyl 1mcgr/kg iv and propofol 1mg/kg iv will be administered to patients for sedation. During the procedure, the BiS value will be arranged 60-85 and propofol 10-30 mg will be administered intravenously if necessary. If sedation is insufficient, fentanyl 25 mcg iv will be added. After baseline values are recorded mean arterial pressure, BiS values, etCO2, RR, SpO2, PR, iPi (Integrated Pulmonary Index) score values will be recorded at 5 minute intervals after the procedure has started. At the end of the procedure, ODI (Oxygenesaturation Index), A/Hr (hourly apnea) values will be recorded.

Undesirable events like apnea, desaturation will be intervened and duration of it will be recorded. Apnea is described as the breathing stops (ETCO2 = 0mmHg, RR = 0 ) for more than 30 seconds and desaturation is described the fall in SpO2 value below 4% of initial value lasting for at least 4 minutes. When apnea and desaturation are seen, verbal stimulation, jaw lifting maneuver and oxygen flow will be increased. If the apnea and desaturation periods of the patients are prolonged or the SpO2 value falls below 10% of the initial value despite the interventions, the procedure will be terminated and necessary procedures will be performed to ensure airway safety and the study will be terminated.

Patients who have completed the endoscopic intervention will be taken to the recovery unit and the Fast-tracking recovery score will be calculated at 10 minute intervals in the first hour. The time that the fast-tracking score is 14 will be recorded. Patients with two consecutive Fast-tracking recovery score values 14 will be discharged. Patients will be called after 24-48 hours and questioned if they have symptoms such as abdominal distension, fever, nausea and vomiting, dizziness and weakness. The satisfaction score to the patient will be questioned; 1:not satisfied at all, 2: not satisfied, 3: neutral, 4:satisfied, 5: very satisfied.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* underwent gastrointestinal endoscopy

Exclusion Criteria:

* existing heart and lung disease
* liver and kidney failure
* morbid obese
* using psychiatric drugs
* having malignancy
* pregnant and lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
early detection of adverse events | 30 minutes
  early detection of adverse events in patients who underwent sedation during gastrointestinal endoscopic intervention in the endoscopy unit

SECONDARY OUTCOMES:
quality of recovery period | 120 minutes
  Fast-tracking recovery score is eveluaed for quality of recovery period
Patients satisfaction | 24 hours
  Patients is called for eveluating for their satisfaction. (1:not satisfied at all, 2: not satisfied, 3: neutral, 4:satisfied, 5: very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Nurten Bakan, doctor, Study Director — Ministry of Health University
Locations (1):
- S.B.U. Sancaktepe Education and Research Hospital, Istanbul, Turkey (Türkiye)